CLINICAL TRIAL: NCT06634901
Title: The Impact of Health Literacy Education on Knowledge, Treatment Adherence and Stigma Among Adolescents With Epilepsy
Brief Title: Health Literacy Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Mbarara Regional Referral Hospital (Unknown); Butabika National Referral Mental Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00116250
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Literacy Educational Session- Control Group Testing (Active Comparator): Participants will receive pre- and post-testing at the same interval as the experimental arm. Rather than receiving the educational session intervention, participants will have lunch during the interval. The comparator group will receive the intervention after all primary and secondary outcome measures have been completed.
  Interventions: Other: Health Literacy Educational Session- Comparator; Behavioral: Health Literacy Educational Session
- Health Literacy Educational Session- Experimental Group Testing (Experimental): Participants are divided into groups of 6-10 adolescents each to receive the educational session intervention, with those aged 12-15 in different groups from those aged 16-18 due to potential differences in question focus.
  Interventions: Behavioral: Health Literacy Educational Session

INTERVENTIONS:
Other: Health Literacy Educational Session- Comparator — During the pre-to-post-test interval for the Knowledge, Attitudes, and Practices (KAP) measure, participants in this arm will take a break and have lunch.
  Arms: Health Literacy Educational Session- Control Group Testing
Behavioral: Health Literacy Educational Session — The Intervention is a 90 minute small group (n=6-10) session with an expert epilepsy provider reviewing fundamental information about epilepsy being a treatable neurologic condition, with topics including epidemiology, causation facts and myths, treatment and the importance of consistent medication, stigma, barriers to care and well-being. These topics will be covered in the first 45 minutes, leaving the second 45 minutes for Q&A with the expert. This session provides the basic health information relevant to people with epilepsy, communication of which is often sacrificed in overcrowded clinics found in low resource settings.

SUMMARY:
Evaluating changes in knowledge, attitude, and practices (KAP) related to epilepsy and its treatment as a result of an educational intervention among adolescents with epilepsy to determine if improved KAP about epilepsy results in improved medication adherence and less perceived stigma.

DETAILED DESCRIPTION:
This proof-of-concept study aims to evaluate the impact of a targeted health literacy intervention on knowledge and attitudes about epilepsy and its treatment, and reported medication adherence and stigma among adolescents with epilepsy in Uganda.

Research Questions:

1. What is the impact of a culturally relevant information session on the knowledge of epilepsy and its treatment among adolescents with epilepsy in Uganda?
2. What is the impact of such an educational session on reported medication adherence and reported stigma among this group?

The investigators hypothesize that a culturally relevant educational intervention will significantly improve knowledge about epilepsy and its treatment, increase medication adherence, and reduce stigma among adolescents with epilepsy in Uganda. This hypothesis is based on the premise that tailored health literacy interventions can address specific misconceptions and barriers to care, thereby improving health outcomes for PWE (persons with epilepsy) in contexts burdened by significant treatment gaps and cultural stigmatization.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a diagnosis of epilepsy attending a clinic at one of the study sites.
* Ages 12-18 years
* Ability and willingness to provide informed assent and guardian consent to participate in the study.
* English, Runyankole or Luganda language proficiency.

Exclusion Criteria:

* Unable or unwilling to provide informed consent or assent to participate in the study.
* Developmental/cognitive challenges that hinder participation in the intervention or completion of surveys.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Epilepsy Knowledge, Attitudes, and Practices (KAP) | 20 minutes
  The primary outcome measure is a 31-item Knowledge, Attitudes, and Practices (KAP) about epilepsy survey. The questionnaire was adapted from Krishnaiah and colleagues (2016), and measures basic knowledge about and attitudes toward epilepsy. Epilepsy Knowledge & Attitudes (KAP) has a reporting scale: 0-31 (higher better).

SECONDARY OUTCOMES:
Kilifi Stigma Scale | 10 minutes
  This 15-item survey was developed and validated in Kilifi, Kenya to measure stigma, and has been used extensively in epilepsy survey research in East Africa. The reporting scale for the Kilifi Stigma Scale: 0-30 (higher worse)
Voils Medication Adherence Items | 3-minutes
  Three items from Voils Medication Adherence (2012) measure will be used to estimate reported medication adherence. The reporting scale for Voil's Medication Adherence: 3-15 (higher worse).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Koltai, MD, Principal Investigator — Duke University
Locations (2):
- Uganda (2):
  - Mayanja Memorial Hospital, Mbarara
  - Mbarara Regional Referral Hospital, Mbarara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biset G, Abebaw N, Gebeyehu NA, Estifanos N, Birrie E, Tegegne KD. Prevalence, incidence, and trends of epilepsy among children and adolescents in Africa: a systematic review and meta-analysis. BMC Public Health. 2024 Mar 12;24(1):771. doi: 10.1186/s12889-024-18236-z. PMID 38475724
- [Background] Meyer AC, Dua T, Ma J, Saxena S, Birbeck G. Global disparities in the epilepsy treatment gap: a systematic review. Bull World Health Organ. 2010 Apr;88(4):260-6. doi: 10.2471/BLT.09.064147. Epub 2009 Sep 25. PMID 20431789
- [Background] Owolabi LF, Owolabi SD, Adamu B, Jibo AM, Alhaji ID. Epilepsy treatment gap in Sub-Saharan Africa: Meta-analysis of community-based studies. Acta Neurol Scand. 2020 Jul;142(1):3-13. doi: 10.1111/ane.13246. Epub 2020 Apr 14. PMID 32219865
- [Background] Kirabira J, Nakawuki M, Fallen R, Zari Rukundo G. Perceived stigma and associated factors among children and adolescents with epilepsy in south western Uganda: A cross sectional study. Seizure. 2018 Apr;57:50-55. doi: 10.1016/j.seizure.2018.03.008. Epub 2018 Mar 8. PMID 29567525
- [Background] Sanchez N, Kajumba M, Kalyegira J, Sinha DD, Bobholz S, Gualtieri A, Chakraborty P, Onuoha E, Fuller AT, Teuwen DE, Haglund MM, Koltai DC. Stakeholder views of the practical and cultural barriers to epilepsy care in Uganda. Epilepsy Behav. 2021 Jan;114(Pt B):107314. doi: 10.1016/j.yebeh.2020.107314. Epub 2020 Aug 3. PMID 32758404
- [Background] Kaddumukasa M, Kaddumukasa MN, Buwembo W, Munabi IG, Blixen C, Lhatoo S, Sewankambo N, Katabira E, Sajatovic M. Epilepsy misconceptions and stigma reduction interventions in sub-Saharan Africa, a systematic review. Epilepsy Behav. 2018 Aug;85:21-27. doi: 10.1016/j.yebeh.2018.04.014. Epub 2018 Jun 13. PMID 29906697
- [Background] Ngugi AK, Kariuki SM, Bottomley C, Kleinschmidt I, Sander JW, Newton CR. Incidence of epilepsy: a systematic review and meta-analysis. Neurology. 2011 Sep 6;77(10):1005-12. doi: 10.1212/WNL.0b013e31822cfc90. PMID 21893672
- [Background] Ba-Diop A, Marin B, Druet-Cabanac M, Ngoungou EB, Newton CR, Preux PM. Epidemiology, causes, and treatment of epilepsy in sub-Saharan Africa. Lancet Neurol. 2014 Oct;13(10):1029-44. doi: 10.1016/S1474-4422(14)70114-0. PMID 25231525
- [Background] Kaddumukasa MN, Kaddumukasa M, Kajumba M, Smith PJ, Bobholz S, Kakooza-Mwesige A, Sinha DD, Almojuela A, Chakraborty P, Nakasujja N, Nakku J, Gualtieri A, Onuoha E, Kolls BJ, Muhumuza C, Smith CE, Sanchez N, Fuller AT, Haglund MM, Koltai DC. Barriers to biomedical care for people with epilepsy in Uganda: A cross-sectional study. Epilepsy Behav. 2021 Jan;114(Pt B):107349. doi: 10.1016/j.yebeh.2020.107349. Epub 2020 Sep 20. PMID 32962922
- [Background] Beghi E. The Epidemiology of Epilepsy. Neuroepidemiology. 2020;54(2):185-191. doi: 10.1159/000503831. Epub 2019 Dec 18. PMID 31852003
- [Background] Scott AJ, Sharpe L, Hunt C, Gandy M. Anxiety and depressive disorders in people with epilepsy: A meta-analysis. Epilepsia. 2017 Jun;58(6):973-982. doi: 10.1111/epi.13769. Epub 2017 May 3. PMID 28470748
- [Background] Adewuya AO, Ola BA. Prevalence of and risk factors for anxiety and depressive disorders in Nigerian adolescents with epilepsy. Epilepsy Behav. 2005 May;6(3):342-7. doi: 10.1016/j.yebeh.2004.12.011. PMID 15820341
- [Background] Mbuba CK, Newton CR. Packages of care for epilepsy in low- and middle-income countries. PLoS Med. 2009 Oct;6(10):e1000162. doi: 10.1371/journal.pmed.1000162. Epub 2009 Oct 13. PMID 19823570
- [Background] Nicholas A. Unlocking the hidden burden of epilepsy in Africa: Understanding the challenges and harnessing opportunities for improved care. Health Sci Rep. 2023 Apr 17;6(4):e1220. doi: 10.1002/hsr2.1220. eCollection 2023 Apr. PMID 37081998
- [Background] Krishnaiah B, Alwar SP, Ranganathan LN. Knowledge, attitude, and practice of people toward epilepsy in a South Indian village. J Neurosci Rural Pract. 2016 Jul-Sep;7(3):374-80. doi: 10.4103/0976-3147.181490. PMID 27365954
- [Background] Mbuba CK, Abubakar A, Odermatt P, Newton CR, Carter JA. Development and validation of the Kilifi Stigma Scale for Epilepsy in Kenya. Epilepsy Behav. 2012 May;24(1):81-5. doi: 10.1016/j.yebeh.2012.02.019. Epub 2012 Apr 4. PMID 22481043
- [Background] Voils CI, Maciejewski ML, Hoyle RH, Reeve BB, Gallagher P, Bryson CL, Yancy WS Jr. Initial validation of a self-report measure of the extent of and reasons for medication nonadherence. Med Care. 2012 Dec;50(12):1013-9. doi: 10.1097/MLR.0b013e318269e121. PMID 22922431
- [Background] Cicero CE, Giuliano L, Todaro V, Colli C, Padilla S, Vilte E, Crespo Gomez EB, Camargo Villarreal WM, Bartoloni A, Zappia M, Nicoletti A. Comic book-based educational program on epilepsy for high-school students: Results from a pilot study in the Gran Chaco region, Bolivia. Epilepsy Behav. 2020 Jun;107:107076. doi: 10.1016/j.yebeh.2020.107076. Epub 2020 Apr 18. PMID 32315969